CLINICAL TRIAL: NCT07038811
Title: Implementation of the App Tät®II for Treatment of Urgency and Mixed Urinary Incontinence
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Region Jämtland Härjedalen (Other)
Responsible Party: Sponsor
Other Study IDs: CIV-24-10-049439
Record Dates: First submitted 2025-06-12; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Urgency Incontinence; Mixed Incontinence, Urge and Stress
Keywords: urinary incontinence; app treatment
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with symptoms of urgency urinary incontinence or mixed urinary incontinence.: Persons of the female gender, aged 18 years or older, with symptoms of urgency urinary incontinence or mixed urinary incontinence, who have undergone a medical evaluation and received a diagnosis of urinary incontinence from a primary care physician.
  Interventions: Device: Tät®II

INTERVENTIONS:
Device: Tät®II — The Tät®II app offers a treatment program for women with urge or mixed urinary incontinence. The program includes information on the pelvic floor, urinary incontinence, and factors affecting incontinence; a bladder training program; a pelvic floor muscle training program; and incontinence-related psychoeducation. The app also contains helpful functions, the ability to create reminders, visualization of each training level, a statistics function regarding the number of exercises performed, and feedback on changes in the level of bother due to urinary incontinence during treatment.
  The Tät®II app is available for download on Google Play and the App Store. Users need a one-time code to access the app, which is provided by the research team after they are included in the study. The app is self-instructive and can be used anywhere; no formal education is necessary. There is no option to communicate through the app.

SUMMARY:
This observational study aims to evaluate the implementation and use of the Tät®II app for the treatment of urgency and mixed urinary incontinence in women over the age of 18 after contact with ordinary healthcare, as well as its effectiveness. The study aims to answer the following question:

Is treatment via the app effective and feasible after primary care?

Participants will use the app for 15 weeks to treat urgency and mixed urinary incontinence. They will answer online survey questions about their urinary incontinence before, after 15 weeks, and one year after treatment.

DETAILED DESCRIPTION:
The implementation study includes women diagnosed with urgency or mixed urinary incontinence by their doctor and recommended first-line treatment with pelvic floor muscle training and/or bladder training.

We plan to recruit eligible participants by advertising in primary care center waiting rooms, on social media, and on our research webpage. Primary care doctors and nurses will also receive information about the study. Women interested in the study from all over Sweden can visit our webpage (tät.nu) for more information. The webpage will include detailed information about the study, the informed consent procedure, an informed consent form, a screening questionnaire, and contact details for the research group.

Women interested in participating in the study are asked to read the subject information and answer the screening questionnaire describing the inclusion and exclusion criteria. Those who are eligible will be asked to send their email address to the research group, which will then contact them by email to schedule a secure video meeting.

During the digital meeting, the investigators will provide additional information about the study and answer any questions. The investigator will also verify that the woman meets all the inclusion criteria and none of the exclusion criteria.

To certify that she has received a medical evaluation for her urinary incontinence, she must send the research team a copy of a medical record. The assessment must not be older than six months.

If she is eligible and wants to participate in the study, she will sign the informed consent form during the meeting and send it to the research group by regular mail. At the same time, she will send a copy of the medical record to the research group as verification of the evaluation.

The investigators will sign the informed consent form as soon as they receive it and then resend a copy to the participant.

Once the informed consent form is signed by both parties, the woman is included in the study.

After inclusion, the research group will send a link to an electronic baseline questionnaire. This questionnaire will include questions about demographics, medical history (including gynecological history and medications), health and eHealth literacy, and validated questionnaires for assessing symptoms and quality of life. The ICIQ-UI SF (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form) and ICIQ-LUTSqol (International Consultation on Incontinence Questionnaire-Lower Urinary Tract Symptoms) validated scores will be used to evaluate symptoms and quality of life.

After completing the questionnaire, participants will have access to the app for 15 weeks of treatment. The research group will email the participants an activation code that can be used to access the app fully.

After 15 weeks and 1 year, a digital follow-up questionnaire will be sent via email. This questionnaire will include validated questionnaires for symptoms (ICIQ-UI SF), quality of life (ICIQ-LUTSqol), and impression of improvement (PGI-I).

The primary outcome for the treatment effect is the validated, widely used ICIQ-UI SF symptom score. A paired t-test will analyze changes in the mean ICIQ-UI SF score from inclusion to follow-up.

Based on the results of the RCT, it is estimated that approximately 60 participants are required. Information on patient experience with app management, satisfaction with management, and desire for further treatment will also be collected. A subgroup analysis will compare the symptoms, effects, and experiences of women 65 years and older to those of women younger than 65.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age ≥18 years
* Symptoms of urgency urinary incontinence or mixed urinary incontinence
* Medical evaluation and documentation of urinary incontinence by ordinary doctor
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Childbirth in the last 6 months
* Painful urges
* Difficulties emptying the bladder
* Blood in urine
* Need of further investigation concerning the urinary incontinence, according to the clinical doctor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women from all over Sweden
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Is treatment via Tät®II effective and feasible after contact with the primary care? | From participants enrollment to the end of treatment at 15 weeks.
  The primary outcome for the treatment effect is the validated and widely used ICIQ-UI SF (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form) symptom score. The ICIQ-UI SF includes three questions about urinary incontinence: how often it occurs, how much leakage there is, and how bothersome it is. These questions form an additive score ranging from 0 to 21 points. The questionnaire also includes a fourth question that is not included in the total score, but that is used to categorize the type of leakage.
  Web-based questionnaires will be sent via email at the beginning of the study and again after 15 weeks. These questionnaires will include the validated ICIQ-UI SF symptom questionnaire.
  Primary endpoint:
  The mean difference in the ICIQ-UI SF score from baseline to the 15-week follow-up.

SECONDARY OUTCOMES:
How does the quality of life (QoL) change after 15 weeks of treatment with the Tät®II app? | From enrollment to the end of treatment at 15 weeks.
  A validated patient-completed questionnaire will be used (International Consultation on Incontinence Questionnarre - Lower Urinary Tract Symtoms (ICIQ-LUTSqol) to evaluate QoL. It contains 20 questions, scoring from 19 to 76, with greater values indicating an increased impact of QoL.
Patient Global Impression of Improvement at 15-week follow up | From enrollment to the end of treatment at 15 weeks.
  A validated patient-completed questionnaire will be used (Patient Global Impression of Improvement scale (PGI-I)) to evaluate improvement. The PGI-I is a single item questionnaire that asks the participant to rate her condition after treatment on a 7 step Likert-scale ranging from "Very much worse" to "Very much better".

CONTACTS AND LOCATIONS:
Overall Officials: Ina Asklund, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Region Jämtland Härjedalen, Östersund, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD directly because the data set is small and contains sensitive information about health conditions. However, the IPD might be shared upon reasonable request.

REFERENCES:
- [Background] Wadensten T, Nystrom E, Sjostrom M, Lindam A, Samuelsson E. APP-based treatment of urgency and mixed urinary incontinence in women: factors associated with long-term satisfaction. Arch Gynecol Obstet. 2024 May;309(5):2193-2202. doi: 10.1007/s00404-023-07303-2. Epub 2023 Dec 23. PMID 38141064
- [Background] Wadensten T, Nystrom E, Nord A, Lindam A, Sjostrom M, Samuelsson E. App-based self-management of urgency and mixed urinary incontinence in women: One-year follow-up. Neurourol Urodyn. 2022 Apr;41(4):945-954. doi: 10.1002/nau.24898. Epub 2022 Mar 9. PMID 35266189
- [Background] Wadensten T, Nystrom E, Franzen K, Lindam A, Wasteson E, Samuelsson E. A Mobile App for Self-management of Urgency and Mixed Urinary Incontinence in Women: Randomized Controlled Trial. J Med Internet Res. 2021 Apr 5;23(4):e19439. doi: 10.2196/19439. PMID 33818395
- See also: Homepage of the research group with information about the study and link to the screening survey. — https://xn--tt-via.nu/